CLINICAL TRIAL: NCT06566716
Title: Validation of Ovarian Adnexal Mass Assessment Score Test System
Brief Title: A Diagnostic Test to Evaluate Cancer Risk Before Surgery in Women with an Ovarian Mass
Status: Recruiting | Type: Observational
Sponsor: Cleo Diagnostics Ltd (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP-01-001
Record Dates: First submitted 2024-08-17; First posted 2024-08-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Neoplasms
Keywords: ovarian; adnexal; benign; malignant; cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Malignant: Patients with an adnexal mass that is surgically diagnosed as malignant
  Interventions: Diagnostic Test: CleoDX ovarian cancer test
- Non-Malignant: Patients with an adnexal mass that is surgically diagnosed as benign
  Interventions: Diagnostic Test: CleoDX ovarian cancer test

INTERVENTIONS:
Diagnostic Test: CleoDX ovarian cancer test — A diagnostic test to assist in predicting risk of malignancy prior to surgery for patients with an adnexal mass.

SUMMARY:
Ovarian cancer is a serious health risk with the highest death rate among gynecological cancers. Unfortunately, it's only possible to definitively diagnose ovarian cancer after surgery, as there are no reliable tests to determine if an ovarian abnormality is cancerous or benign before surgery.

Cleo Diagnostics have developed a new test that uses five biomarkers in the blood to better differentiate between benign and malignant ovarian conditions. In initial studies, this test outperformed the current standard test, CA125, in identifying cancer.

This study aims to evaluate the effectiveness of the Cleo Diagnostics (CleoDX) Ovarian Adnexal Mass Score Test System. This test measures five analytes in the blood and provides a score indicating the likelihood of cancer in patients with an adnexal mass requiring surgery. The test is designed to assist doctors in making better-informed decisions about surgery and patient care by providing a more accurate pre-surgical assessment of cancer risk. By doing so, it aims to improve patient outcomes and ensure that those with malignant conditions receive the appropriate specialist care.

ELIGIBILITY:
Inclusion Criteria:

* female patients => 18 years of age at the time of consent
* Can provide written informed consent
* Have an ovarian cyst or adnexal mass (simple, complex, or solid ovarian/pelvic mass) identified through imaging examination (e.g. transvaginal ultrasound - TVU) that requires surgery, but have not yet undergone this surgery

Exclusion Criteria:

* Any prior confirmed diagnosis of, or treatment for, ovarian cancer
* Any prior surgery resulting in removal of both ovaries
* Prior history of gynecological malignancy (within last 2 years)
* Prior history of melanoma (within last 2 years)
* Prior treatment (within 12 months of sample collection) with chemotherapy, radiotherapy or immunotherapy
* Immune-compromised. Definition: those whose weakened immune system may render them more susceptible to infection, illness, or complications. These may include patients with immune-suppressive conditions (e.g. HIV/AIDS), patients undergoing immuno-, chemo- or radio-therapy (within the last 12 months) for any reason, receiving immune suppressive therapies (e.g. transplant recipients, individuals with known autoimmune disease), or with a primary immunodeficiency disorder (e.g. Lupus).
* Pregnant currently or within the last 3 months based on participant self-report

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants identified at general medical clinics and hospital in-patient gynecology clinics with visible ovarian or pelvic abnormality on ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Calculation of the CleoDX adnexal mass score | Outcomes will be assessed during an analysis phase, which will commence after completion of patient recruitment and continue for up to 12 months or the end of the study period is reached (August 2026), whichever occurs first.
  Determine the Cleo Diagnostics (CleoDX) adnexal mass score in patients identified with an adnexal mass requiring surgery, but who have not yet undergone this surgery.

SECONDARY OUTCOMES:
Compare CleoDX adnexal mass score with pre- and post-surgical clinicopathologic information | Outcomes will be assessed during an analysis phase, which will commence after completion of patient recruitment and continue for up to 12 months or the end of the study period is reached (August 2026), whichever occurs first.
  Correlate post-surgical pathology findings with the CleoDX adnexal mass score, and evaluate the performance metrics (including sensitivity, specificity, Negative Predictive Value and Positive Predictive Value) of the CleoDX adnexal mass assessment scoring system.
Determine performance and accuracy of the CleoDX test against post-surgical pathology findings | Outcomes will be assessed during an analysis phase, which will commence after completion of patient recruitment and continue for up to 12 months or the end of the study period is reached (August 2026), whichever occurs first.
  Correlate post-surgical pathology findings with the CleoDX adnexal mass score, and evaluate the performance metrics (including sensitivity, specificity, Negative Predictive Value and Positive Predictive Value) of the CleoDX adnexal mass assessment scoring system.
Identify rate of accurately predicted diagnoses by CleoDX compared to that of standard clinical workflow | Outcomes will be assessed during an analysis phase, which will commence after completion of patient recruitment and continue for up to 12 months or the end of the study period is reached (August 2026), whichever occurs first.
  Demonstrate superiority of the CleoDX adnexal mass scoring system compared to standard clinical workflows including CA125 and Risk of Malignancy Index (RMI) measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Director — Cleo Diagnostics Ltd
Locations (8):
- United States (8):
  - New Horizons Clinical Trials, Chandler, Arizona
  - Emerald Coast Clinical Research, Panama City, Florida
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - The Jackson Clinic, Jackson, Tennessee
  - Next Innovative Clinical Research, Houston, Texas
  - Prime Clinical Research - Lewisville, Lewisville, Texas
  - Vast Clinical Research-Holy Cross, Mesquite, Texas
  - Virginia Women's Health Associates, Annandale, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stephens AN, Hobbs SJ, Kang SW, Bilandzic M, Rainczuk A, Oehler MK, Jobling TW, Plebanski M, Allman R. A Novel Predictive Multi-Marker Test for the Pre-Surgical Identification of Ovarian Cancer. Cancers (Basel). 2023 Nov 2;15(21):5267. doi: 10.3390/cancers15215267. PMID 37958440
- [Background] Stephens AN, Hobbs SJ, Kang SW, Oehler MK, Jobling TW, Allman R. Utility of a Multi-Marker Panel with Ultrasound for Enhanced Classification of Adnexal Mass. Cancers (Basel). 2024 May 28;16(11):2048. doi: 10.3390/cancers16112048. PMID 38893167
- [Background] Stephens AN, Hobbs SJ, Kang SW, Oehler MK, Jobling TW, Allman R. ReClassification of Patients with Ambiguous CA125 for Optimised Pre-Surgical Triage. Diagnostics (Basel). 2024 Mar 22;14(7):671. doi: 10.3390/diagnostics14070671. PMID 38611584